CLINICAL TRIAL: NCT03052088
Title: A Multi-center, Prospective, Pilot Study to Validate the Diagnostic Accuracy and Assess the Potential Clinical Utility of a Host-response Based Diagnostic Tool for Distinguishing Between Bacterial and Viral Etiologies in Pediatric Patients Presenting to the Emergency Department With Respiratory Tract Infection (RTI) or Fever Without Source (FWS)
Brief Title: Diagnostic Accuracy of a Host-response Based Diagnostic Tool for Distinguishing Between Bacterial and Viral Etiologies in Pediatric Patients
Acronym: AutoPilot
Status: Completed | Type: Observational
Sponsor: MeMed Diagnostics Ltd. (Industry)
Collaborators: European Commission (Other); Heidelberg University (Other); University of Parma (Other)
Responsible Party: Sponsor
Other Study IDs: MM-1006-AP
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Fever; Respiratory Tract Infections
MeSH Terms: conditions — Fever; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective clinical validation study of a novel regulatory approved (CE-IVD) diagnostic assay called ImmunoXpert™ that will enroll 1222 pediatric patients. The study aims to externally validate the tool's diagnostic accuracy and estimate the potential improvement in health and economic outcomes following the usage of ImmunoXpert™. Additionally, statistical analysis will be performed to compare ImmunoXpert™ accuracy to current practice lab testing (e.g. WBC, CRP, and PCT) and clinical suspicion at time of requisition. Enrolled patients will be managed according to the current standard of care and per standard institutional procedures.

ELIGIBILITY:
Inclusion Criteria:

* Legal guardian signs an informed consent
* Documented peak temperature ≥ 38°C (100.4°F)
* Symptom duration ≤ 7 days
* Clinical suspicion of RTI (OR) fever without a clear source after clinical examination

Exclusion Criteria:

* Another episode of febrile infection within the past 2 weeks
* Antibiotic treatment of over 48 hours
* Congenital immune deficiency (CID)
* A proven or suspected HIV, HBV, HCV infection
* Active malignancy
* Current treatment with immune-suppressive or immune-modulating therapies, including without limitations:
* Use of high dose steroids >1 mg/kg/day prednisone or equivalent in the past two weeks
* Monoclonal antibodies, anti-TNF agents
* Intravenous immunoglobulin (IVIG)
* Cyclosporine, Cyclophosphamide, Tacrolimus
* G/GM-CSF, Interferons
* Other severe illnesses that affect life expectancy and/or quality of life such as:
* Severe psychomotor retardation
* Post-transplant patients
* Severe congential metabolic disorder

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible subjects from both genders that present to the ED due to suspected RTI, or FWS. Each of these patients falls into one of the following categories:
  1. Patients with an acute bacterial infection
  2. Patients with an acute viral infection
  3. Patients with an acute co-infection (bacterial and viral)
  4. Patients with an undetermined disease etiology
Sampling Method: Probability Sample
Enrollment: 1140 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
To validate the diagnostic accuracy and assess the clinical utility of a host-response based diagnostic tool, for differentiating between bacterial and viral etiologies in pediatric patients >90 days old with suspicion of RTI or FWS | 0-7 days after the initiation of symptoms

SECONDARY OUTCOMES:
To compare the diagnostic accuracy of a host-response based diagnostic to currently available lab measures (WBC, ANC, CRP and PCT), using sensitivity and specificity measures and predetermined cutoffs | 0-7 days after the initiation of symptoms
To compare ImmunoXpert™ results with the physician suspected diagnosis at time of patient recruitment and compared to the reference standard diagnosis | 0-7 days after the initiation of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Tenenbaum, MD, Principal Investigator — Kinderklinik Universitatsmedizine mannheim
Locations (2):
- Kinderklinik Universitatsmedizin Mannheim, Mannheim, Germany
- Pietro Barilla Children's Hospital, Parma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oved K, Cohen A, Boico O, Navon R, Friedman T, Etshtein L, Kriger O, Bamberger E, Fonar Y, Yacobov R, Wolchinsky R, Denkberg G, Dotan Y, Hochberg A, Reiter Y, Grupper M, Srugo I, Feigin P, Gorfine M, Chistyakov I, Dagan R, Klein A, Potasman I, Eden E. A novel host-proteome signature for distinguishing between acute bacterial and viral infections. PLoS One. 2015 Mar 18;10(3):e0120012. doi: 10.1371/journal.pone.0120012. eCollection 2015. PMID 25785720
- [Background] Eden E, Srugo I, Gottlieb T, Navon R, Boico O, Cohen A, Bamberger E, Klein A, Oved K. Diagnostic accuracy of a TRAIL, IP-10 and CRP combination for discriminating bacterial and viral etiologies at the Emergency Department. J Infect. 2016 Aug;73(2):177-80. doi: 10.1016/j.jinf.2016.05.002. Epub 2016 May 30. No abstract available. PMID 27255416
- [Background] van Houten CB, de Groot JAH, Klein A, Srugo I, Chistyakov I, de Waal W, Meijssen CB, Avis W, Wolfs TFW, Shachor-Meyouhas Y, Stein M, Sanders EAM, Bont LJ. A host-protein based assay to differentiate between bacterial and viral infections in preschool children (OPPORTUNITY): a double-blind, multicentre, validation study. Lancet Infect Dis. 2017 Apr;17(4):431-440. doi: 10.1016/S1473-3099(16)30519-9. Epub 2016 Dec 22. PMID 28012942